CLINICAL TRIAL: NCT05128227
Title: PHARM-S.A.V.E.S: Suicide Prevention Gatekeeper Training for Pharmacy Staff
Brief Title: PHARM-S.A.V.E.S: Suicide Prevention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Foundation for Suicide Prevention (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 21-1062
Record Dates: First submitted 2021-10-28; First posted 2021-11-19 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Suicide
Keywords: community pharmacy; communication; gatekeeper training; suicide prevention; pharmacy
MeSH Terms: conditions — Suicide; Communication; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharm-SAVES (Active Comparator): This is an approximately 30-minute self-guided online module that covers basic information about suicide prevention gatekeeper skills training that is relevant to community pharmacists.
  Interventions: Behavioral: Pharm-SAVES
- Interactive video case (Experimental): An approximately 30-minute self-guided online suicide prevention gatekeeper skills training module, plus two approximately 5-minute interactive video cases in which participants are asked to respond to patients who exhibit suicidal warning signs.
  Interventions: Behavioral: Pharm-SAVES; Behavioral: Interactive video cases

INTERVENTIONS:
Behavioral: Pharm-SAVES — A 30 minute long online module with videos and didactic content that covers the following topics: warning signs of suicide, how to ask a patient if they are contemplating suicide, and how to refer a patient to the Crisis Line. Three videos model patient scenarios of suicidal behavior in pharmacy settings including the pharmacy drive through, over the phone, and in person. Participants will receive continuing education credits (CEUs) (0.1 CEUs) for completing the course.
Behavioral: Interactive video cases — Two video interactive cases (approximately 10-minutes combined total) ask participants to complete open and close-ended questions about patients who exhibit suicidal behavior at the pharmacy. Participants will receive continuing education credits (0.1 CEUs) for completing the course.
  Arms: Interactive video case

SUMMARY:
This is a pilot Randomized Controlled Trial (RCT) in which 150 pharmacy staff members will be randomized to an experimental or control group and data on suicide prevention communication and secondary outcomes will be collected over the course of the RCT.

DETAILED DESCRIPTION:
This is a prospective pilot RCT that will evaluate the impact of suicide prevention gatekeeper training (Pharm-SAVES) on 150 pharmacy staff member communication behaviors (primary outcome). Data will be collected at baseline, immediately after training is completed, and at 1-month follow up. Data sources include simulated patient observations (to rate quality of communication) and survey data (for self-reports of knowledge, self-efficacy, and referral behaviors).

ELIGIBILITY:
Inclusion Criteria:

Staff must:

* be at least 18 years of age;
* read and speak English; and
* be currently employed as a pharmacist or pharmacy technician at a community pharmacy

Exclusion Criteria:

* Individuals will be excluded if they hold floater status (non-staff pharmacists or technicians).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in proportion of participants who ask about suicide. | Baseline and immediately post-intervention
  An online survey will include a written case that asks participants what they would say to a patient who has expressed verbal suicide warning sign(s). Blinded coders will review the open-ended response to determine whether the participant asks about suicide. The responses will be coded as no=0 and yes=1.

SECONDARY OUTCOMES:
Change in proportion of participants who report they would call the National Suicide Prevention Lifeline. | Baseline and immediately post-intervention
  An online survey will include a written case with an open-ended question that asks if, and where, participants would refer a patient who has expressed verbal suicide warning sign(s). Blinded coders will review the open-ended response to determine whether the participant reported they would call the National Suicide Prevention Lifeline. The responses will be coded as no=0 and yes=1.
Change in suicide prevention knowledge score from baseline to immediate post-intervention. | Baseline and immediately post-intervention
  An online survey including 5 multiple choice and 5 true-false questions will assess participants suicide prevention knowledge based on the content of Pharm-SAVES.A summary score that assesses the total number of correct answers (range: 0-10) will be created, with higher scores reflecting higher knowledge.
Change in mean suicide prevention self-efficacy score from baseline to immediate post-intervention. | Baseline and immediately post-intervention
  A 6-item scale will be used to assess gatekeeper efficacy, or how confident trainees are that they can perform various suicide prevention tasks, including identifying signs of suicide and making a referral. Response options range from 1=not at all confident to 5=extremely confident. Item responses for each individual will be averaged to create a mean score, with higher scores indicating higher gatekeeper efficacy. Scores will range from 1 to 5.
Change in mean suicide prevention self-efficacy score from baseline to 1-month follow-up | Baseline and 1-month follow-up
  A 6-item scale to will be used assess gatekeeper efficacy, or how confident trainees are that they can perform various suicide prevention tasks, including identifying signs of suicide and making a referral. Response options range from 1=not at all confident to 5=extremely confident. Item responses for each individual will be averaged to create a mean score, with higher scores indicating higher gatekeeper efficacy. Scores will range from 1 to 5.
Change in mean suicide prevention preparedness score from baseline to immediate post-intervention. | Baseline and immediately post-intervention
  Six items from a validated scale will be used to assess gatekeeper preparedness, or how well-prepared trainees feel they are to perform gatekeeper activities, including to "ask appropriate questions about suicide." Response options range from 1=not prepared to 7=quite well-prepared. Item responses for each individual will be averaged, and higher scores will indicate higher levels of gatekeeper preparedness. Scores will range from 1 to 7.
Change in mean suicide prevention preparedness score from baseline to 1-month follow-up. | Baseline and 1-month follow-up
  Six items from a validated scale will be used to assess gatekeeper preparedness, or how well-prepared trainees feel they are to perform gatekeeper activities, including to "ask appropriate questions about suicide." Response options range from 1=not prepared to 7=quite well-prepared. Item responses for each individual will be averaged, and higher scores will indicate higher levels of gatekeeper preparedness. Scores will range from 1 to 7.
Proportion of participants who ask about suicide (optional) | 1-month follow-up
  At 1-month follow-up, participants can choose to complete a video-recorded standardized patient assessment via Zoom. One live standardized patient will enact a scenario in which they express verbal suicide warnings signs. After completion of the live standardized patient (SP) assessment, the participant will watch a pre-recorded video of a second standardized patient who also expressed suicide warning signs. The live SP will then ask the participant how they would respond to the person depicted in the pre-recorded video. Using an observation guide, two masked coders will independently view the videos from each SP scenario and document whether the participant asked a direct question about suicide (yes/no). Examples of direct questions are provided in the observation guide. Scores for asking will range from 0 to 2.

CONTACTS AND LOCATIONS:
Overall Officials: Delesha M Carpenter, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Jill E Lavigne, PhD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF, Analytic Code

REFERENCES:
- [Background] Wyman PA, Brown CH, Inman J, Cross W, Schmeelk-Cone K, Guo J, Pena JB. Randomized trial of a gatekeeper program for suicide prevention: 1-year impact on secondary school staff. J Consult Clin Psychol. 2008 Feb;76(1):104-15. doi: 10.1037/0022-006X.76.1.104. PMID 18229988

DOCUMENTS (1):
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT05128227/ICF_000.pdf